CLINICAL TRIAL: NCT00931476
Title: A Single-centre, Randomised, Double-blind, Placebo-controlled, Parallel Group, Single Dose Trial in Healthy Caucasians and Japanese Subjects Investigating the Pharmacokinetics of Norditropin® (Norditropin® PenSet® 24)
Brief Title: A Single Dose Trial in Healthy Caucasians and Japanese Subjects Investigating the Pharmacokinetics of Somatropin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GHKIN-1253
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency; Healthy
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: somatropin
Drug: placebo

SUMMARY:
This trial was conducted in the United States of America (USA). The aim of this clinical trial was to investigate the pharmacokinetics of somatropin in healthy Japanese and Caucasian subjects, and to identify somatostatin-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent before any trial related activities
* Japanese and Caucasian males respectively
* Healthy subjects based upon medical history, physical examination, vital signs, ECG, serum biochemistry and haematology and urinalysis
* Body Mass Index (BMI) between 17 and 30 m2/kg, inclusive

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2000-04-06 (Actual); Primary Completion 2000-06-08 (Actual); Study Completion 2000-06-08 (Actual)

PRIMARY OUTCOMES:
Area under the hGH concentration-time curve (GH AUC0-24h) | from 0 to 24 hours following injection
Maximum hGH concentration (GH Cmax) | from 0 to 24 hours following injection
Treatment Emergent Adverse Events | from 0 to 24 hours following injection

SECONDARY OUTCOMES:
Time to maximum hGH concentration (GH tmax)
Area under the hGH concentration-time curve GH AUC0-∞)
Elimination half-life (GH t½)
Growth Factors (IGF-I and IGFBP-3)
Non-treatment Emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Honolulu, Hawaii, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com